CLINICAL TRIAL: NCT02341001
Title: Does Text Message Support After Discharge Improve Outcomes Following Bariatric Surgery? A Randomised Trial and Sub-study of the BOBS Study (Better Outcomes Following Bariatric Surgery)
Brief Title: Does Text Message Support After Discharge Improve Outcomes Following Bariatric Surgery? A Randomised Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Collaborators: Health Research Council, New Zealand (Other)
Responsible Party: Principal Investigator, Andrew MacCormick, Senior Lecturer, University of Auckland, New Zealand
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BOBSRCT01
Record Dates: First submitted 2014-11-24; First posted 2015-01-19 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Obesity; Bariatric Surgery Candidate
Keywords: Bariatric surgery; Sleeve gastrectomy; Text messaging; Weight loss; BAROS; Follow-up care
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care (No Intervention): Patients are discharged from the bariatric service at 18 months after surgery.
- Standard care with text message support (Experimental): Patients are discharged from the bariatric service at 18 months after surgery but receive a daily text message for one year.
  Interventions: Other: Daily text message of support

INTERVENTIONS:
Other: Daily text message of support
  Arms: Standard care with text message support

SUMMARY:
The purpose of this study is to determine whether text message support after discharge from a bariatric service improves outcomes following bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have had a sleeve gastrectomy 18 months ago and are attending the discharge follow-up appointment

Exclusion Criteria:

* Patients who do not have the ability to receive text messages
* Patients who do not understand written English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-01; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Percent of excess weight lost | Twelve months

SECONDARY OUTCOMES:
Bariatric Analysis and Reporting Outcome System (BAROS) | Twelve months

OTHER OUTCOMES:
Number of re-referrals to the bariatric clinic | Twelve months
Cost comparison | Twelve months
  Very basic cost comparison will be performed by calculating the cost of each intervention and comparing them. Items included in the cost analysis will be the cost of text messaging and the costs incurred if patients in the study were reviewed by the bariatric team after re-referral.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D MacCormick, MBChB, PhD, Principal Investigator — University of Auckland, New Zealand; Melanie Lauti, MBChB, Principal Investigator — University of Auckland, New Zealand
Locations (1):
- Counties Manukau District Health Board, Auckland, New Zealand

REFERENCES:
- [Derived] Lauti M, Kularatna M, Pillai A, Hill AG, MacCormick AD. A Randomised Trial of Text Message Support for Reducing Weight Regain Following Sleeve Gastrectomy. Obes Surg. 2018 Aug;28(8):2178-2186. doi: 10.1007/s11695-018-3176-1. PMID 29500678